CLINICAL TRIAL: NCT03455465
Title: Using Rapid Cycle Trials to Increase Patient Engagement in the Community Health Worker Program in the Emergency Department at NYU Langone Health Hospital-Brooklyn
Brief Title: Using Rapid Cycle Trials to Increase Patient Engagement in the Community Health Worker Program in the Emergency Department
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-CHW
Record Dates: First submitted 2018-02-14; First posted 2018-03-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Patient Engagement; Community Health Workers
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No intervention: Patients in this arm will not be approached by community health workers during their visit to the Emergency Department.
- Community Health Worker Program: Participants in this group will be approached by a community health worker during their visit to the Emergency Department with the goal of enrolling them in a comprehensive post-discharge program.
  Interventions: Other: Community Health Worker Assessment

INTERVENTIONS:
Other: Community Health Worker Assessment — Participants will be approached by a community health worker who will ask them to complete an assessment of needs and offer to enroll them in post-discharge services to help address the needs identified.
  Groups: Community Health Worker Program

SUMMARY:
This study is evaluating the effectiveness of the post-discharge program facilitated by the Community Health Worker program in the Emergency Department at NYU Langone Health Hospital - Brooklyn and testing different strategies to increase patient engagement in the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present for a visit at the Emergency Department at NYU Langone Brooklyn Hospital and who qualify for the Community Health Worker program assessment and enrollment.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present for a visit at the Emergency Department at NYU Langone Brooklyn Hospital and who qualify for the Community Health Worker program assessment and enrollment.
Sampling Method: Probability Sample
Enrollment: 2314 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Service utilization | 1 year
  Number of services (emergency department visits, etc.) utilized by the patient.
Post-discharge program enrollment rate | 1 year
  Total number of patients who agree to enroll in the post-discharge program/total number of patients approached by community health workers.

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided